CLINICAL TRIAL: NCT05051501
Title: Biotechnology Research Into Microbiological Spectrum Changes to Improve Cognitive Functions, Depression and Other Neuropsychiatric Disorders in Aging Population
Brief Title: The Effects of Microbiological Spectrum Changes to Improve Cognitive Health in Aging Population
Acronym: CleverAgeBiota
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health, Czech Republic (Other)
Collaborators: C2P s.r.o. (Unknown); University Hospital Vinohrady (Unknown); Ministry of Industry and Trade, Czech Republic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: FV-40032
Record Dates: First submitted 2021-04-28; First posted 2021-09-21 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Memory Deficits; Mood Change; Gut Health; Aging Problems; Aging; Cognitive Decline
Keywords: Probiotics; Microbiome; Gut Microflora; Cognitive Health
MeSH Terms: conditions — Memory Disorders; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: First 3 months: group A on probiotics; group B on placebo Next 3 months: group A on placebo; group B on probiotics. Next 3 months: no intervention in either group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants with an odd identification number will receive substance A in the first three months and a complementary substance B in the following three months. Participants with an even identification number will receive substance B in the first three months and a complementary substance A in the following three months. Manufacturer of the new probiotics C2P will mark one set of substances as set A and a complementary set of substances as set B. If substance A/B is a probiotic or placebo will be known to a manufacturer only. Investigators and participants are blinded to this information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics C2P/Placebo (Experimental): Crossover design does not confine one group of patients strictly either to an intervention in question or a placebo. Each group will receive both placebo and probiotics in tandem, but in a reversed order.
  Interventions: Dietary Supplement: Probiotics C2P
- Placebo/Probiotics C2P (Experimental): Crossover design does not confine one group of patients strictly either to an intervention in question or a placebo. Each group will receive both placebo and probiotics in tandem, but in a reversed order.
  Interventions: Dietary Supplement: Probiotics C2P

INTERVENTIONS:
Dietary Supplement: Probiotics C2P — Probiotics will supplement normal diet. Unlike other products available on the market, which are usually of bovine origin, our probiotic has been manufactured using human-stemmed lines. The supplements are composed of a mixture of naturally occurring human gut bacteria.

SUMMARY:
The goal of this project is to develop probiotic dietary supplements intended for the elderly, which can modify the composition of the intestinal microbiota typically occurring in the aging population. According to currently held scientific knowledge, it is postulated that the probiotics-induced normalization of the physiological axis in the brain-intestinal microbiota affects the activity of the nervous system. Thus, normalization of this axis should lead to observable improvements in cognitive functions and quality of life.

DETAILED DESCRIPTION:
With an increasing age of the population, the incidence of age-related problems, such as memory deficits or negative changes in mood, is on the rise. On this account, an increased emphasis has been placed on identifying natural ways to reduce the occurrence of such problems. One of the proposed methods to achieve this is to modify the composition of gut bacteria and their by-products, which has shown a surprising, yet highly promising potential to benefit the brain function and blood composition.

In the recent years, gut bacteria have been of great interest to many medical professionals from various disciplines. It is postulated that they might exert some influence on memory and emotions, but there is a lack of evidence to confirm these hypotheses. Our study would like to address this issue and examine the beneficial effects of probiotics into more depth. Probiotics are dietary supplements in the form of bacteria, which are often artificially added e.g. into some dairy products. This is done to promote gut health and to improve the quality of gut microflora.

The subject selection and assessment are summarised as follows: Participants will be pre-selected electronically and given an electronic memory test. Further selection of eligible subjects based on their preliminary results will be followed by the first personal appointment, where each participant will undergo memory and mood-focused psychological testing and testing for gut bacteria composition. One week after the initial appointment, participants will be asked to bring in a stool and urine sample, their blood will be collected and their fitness and dietary habits assessed. Each participant will also be given an electronic watch, which will monitor their physical activity, and supplements in the pill form, which either contain specially cultivated human gut bacteria (i.e. probiotics) or placebo. Identical tests and blood, urine and stool collection will be repeated three months after administering the first pill. The participants will receive another set of pills, which will contain the probiotics if the participant has initially received placebo and vice versa. After three more months, participants will be subjected to the same tests as in the previous two instants. To test for lasting effects of treatment, participants will be tested again after 3 more months and the project will reach its termination.

Using the above-mentioned methods, the aim of this project is to provide sufficient evidence of the beneficial effects of the new probiotics on memory, mood and the biochemical components contained in the blood, stool and urine in elderly population.

ELIGIBILITY:
Inclusion Criteria:

* is 55-80 years of age
* His/her native language is Czech
* Is willing to visit the testing centre four times within half a year
* Is willing to provide blood, urine and stool samples three times within half a year
* Is willing to self-administer the probiotic/placebo pill once every day for half a year
* is self-sufficient (handling finances, travelling without a chaperone, administration of medication, correct phone usage, filling forms, meal preparation)
* Has good vision; Can read and write, glasses are acceptable
* Has good hearing to hear and understand all instructions during examination
* Can walk well (walking aids are acceptable) to attend all the examinations

Exclusion Criteria:

* Suffers with disorder(s) of digestive system, primarily gastrointestinal disorders (celiac disease, ulcerative colitis, Crohn's disease, frequent diarrhoea)
* Had severe neurological difficulties (epilepsy, stroke, severe head trauma, meningitis in the past 10 years, brain surgery, brain tumour, prolonged period(s) in an unconscious state - excluding general anaesthesia)
* Had been treated/Is currently being treated for the following psychiatric disorders: alcohol/medication/drug of abuse dependance, schizophrenia, psychotic disorder, bipolar disorder
* Is taking medication for depression or low mood
* Suffers from internal organ failure (heart, liver or kidney failure etc.)
* Suffered from an oncological problem (cancer) in the past 5 years
* Underwent radiotherapy or chemotherapy in the past
* Underwent a surgery/procedure under general anaesthesia in the past three years or has a planned procedure/surgery under general anaesthesia in the next 6 months over the course of this trial
* Suffered from hepatitis (hepatitis B, C), HIV or syphilis in the past
* Had taken any probiotics in the past three months

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline cognitive function in the Amnesia Light and Brief Assessment (ALBA) at 3 months | baseline to 3 months
  ALBA is a validated measure assessing memory. The scale spans 0-12 points with higher number of points signifying better outcome
Change from baseline cognitive function in the Amnesia Light and Brief Assessment (ALBA) at 6 months | baseline to 6 months
  ALBA is a validated measure assessing memory. The scale spans 0-12 points with higher number of points signifying better outcome
Change from 3 months cognitive function in the Amnesia Light and Brief Assessment (ALBA) at 6 months | 3 months to 6 months
  ALBA is a validated measure assessing memory. The scale spans 0-12 points with higher number of points signifying better outcome
Change from 6 months cognitive function in the Amnesia Light and Brief Assessment (ALBA) at 9 months | 6 months to 9 months
  ALBA is a validated measure assessing memory. The scale spans 0-12 points with higher number of points signifying better outcome
Difference in cognitive function in the Amnesia Light and Brief Assessment (ALBA) at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  ALBA is a validated measure assessing memory. The scale spans 0-12 points with higher number of points signifying better outcome
Difference in cognitive function in the Amnesia Light and Brief Assessment (ALBA) at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  ALBA is a validated measure assessing memory. The scale spans 0-12 points with higher number of points signifying better outcome
Change from baseline cognitive function in the Assessment Battery of Cognition (ABACO) at 3 months | baseline to 3 months
  ABACO is a measure of cognitive function, results are in points and range from 0-35, higher point attainment signals better outcome
Change from baseline cognitive function in the Assessment Battery of Cognition (ABACO) at 6 months | baseline to 6 months
  ABACO is a measure of cognitive function, results are in points and range from 0-35, higher point attainment signals better outcome
Change from 3 months cognitive function in the Assessment Battery of Cognition (ABACO) at 6 months | 3 months to 6 months
  ABACO is a measure of cognitive function, results are in points and range from 0-35, higher point attainment signals better outcome
Change from 6 months cognitive function in the Assessment Battery of Cognition (ABACO) at 9 months | 6 months to 9 months
  ABACO is a measure of cognitive function, results are in points and range from 0-35, higher point attainment signals better outcome
Difference in cognitive function in the Assessment Battery of Cognition (ABACO) at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  ABACO is a measure of cognitive function, results are in points and range from 0-35, higher point attainment signals better outcome
Difference in cognitive function in the Assessment Battery of Cognition (ABACO) at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  ABACO is a measure of cognitive function, results are in points and range from 0-35, higher point attainment signals better outcome
Change from baseline cognitive function in Semantic word recollection (category: animals, 1 min) at 3 months | baseline to 3 months
  Semantic word recollection is a measure of cognitive function, results range from 0-cca 40, more points signify better outcome
Change from baseline cognitive function in Semantic word recollection (category: animals, 1 min) at 6 months | baseline to 6 months
  Semantic word recollection is a measure of cognitive function, results range from 0-cca 40, more points signify better outcome
Change from 3 months cognitive function in Semantic word recollection (category: animals, 1 min) at 6 months | 3 months to 6 months
  Semantic word recollection is a measure of cognitive function, results range from 0-cca 40, more points signify better outcome
Change from 6 months cognitive function in Semantic word recollection (category: animals, 1 min) at 9 months | 6 months to 9 months
  Semantic word recollection is a measure of cognitive function, results range from 0-cca 40, more points signify better outcome
Difference in cognitive function in Semantic word recollection (category: animals, 1 min) at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  Semantic word recollection is a measure of cognitive function, results range from 0-cca 40, more points signify better outcome
Difference in cognitive function in Semantic word recollection (category: animals, 1 min) at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  Semantic word recollection is a measure of cognitive function, results range from 0-cca 40, more points signify better outcome
Change from baseline cognitive function in Rey Auditory Verbal Learning Test (RAVLT) at 3 months | baseline to 3 months
  RAVLT is a validated measure of cognitive function, it has 8 subscales, each of them ranging from 0-15, measured in raw scores which are connected to age-dependent population norm
Change from baseline cognitive function in Rey Auditory Verbal Learning Test (RAVLT) at 6 months | baseline to 6 months
  RAVLT is a validated measure of cognitive function, it has 8 subscales, each of them ranging from 0-15, measured in raw scores which are connected to age-dependent population norm
Change from 3 months cognitive function in Rey Auditory Verbal Learning Test (RAVLT) at 6 months | 3 months to 6 months
  RAVLT is a validated measure of cognitive function, it has 8 subscales, each of them ranging from 0-15, measured in raw scores which are connected to age-dependent population norm
Change from 6 months cognitive function in Rey Auditory Verbal Learning Test (RAVLT) at 9 months | 6 months to 9 months
  RAVLT is a validated measure of cognitive function, it has 8 subscales, each of them ranging from 0-15, measured in raw scores which are connected to age-dependent population norm
Difference in cognitive function in Rey Auditory Verbal Learning Test (RAVLT) at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  RAVLT is a validated measure of cognitive function, it has 8 subscales, each of them ranging from 0-15, measured in raw scores which are connected to age-dependent population norm
Difference in cognitive function in Rey Auditory Verbal Learning Test (RAVLT) at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  RAVLT is a validated measure of cognitive function, it has 8 subscales, each of them ranging from 0-15, measured in raw scores which are connected to age-dependent population norm
Change in baseline cognitive function in Wechsler Adult Intelligence Scale, Third edition (WAIS III) - "Symbols" subtest at 3 months | baseline to 3 months
  The WAIS III, subtest "Symbols" is a validated measure of cognitive function, the point scale ranges from 0-133 with larger point attainment signalling better outcome
Change in baseline cognitive function in Wechsler Adult Intelligence Scale, Third edition (WAIS III) - "Symbols" subtest at 6 months | baseline to 6 months
  The WAIS III, subtest "Symbols" is a validated measure of cognitive function, the point scale ranges from 0-133 with larger point attainment signalling better outcome
Change in 3 month cognitive function in Wechsler Adult Intelligence Scale, Third edition (WAIS III) - "Symbols" subtest at 6 months | 3 months to 6 months
  The WAIS III, subtest "Symbols" is a validated measure of cognitive function, the point scale ranges from 0-133 with larger point attainment signalling better outcome
Change in 6 month cognitive function in Wechsler Adult Intelligence Scale, Third edition (WAIS III) - "Symbols" subtest at 9 months | 6 months to 9 months
  The WAIS III, subtest "Symbols" is a validated measure of cognitive function, the point scale ranges from 0-133 with larger point attainment signalling better outcome
Difference in cognitive function in Wechsler Adult Intelligence Scale, Third edition (WAIS III) - "Symbols" subtest at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  The WAIS III, subtest "Symbols" is a validated measure of cognitive function, the point scale ranges from 0-133 with larger point attainment signalling better outcome
Difference in cognitive function in Wechsler Adult Intelligence Scale, Third edition (WAIS III) - "Symbols" subtest at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  The WAIS III, subtest "Symbols" is a validated measure of cognitive function, the point scale ranges from 0-133 with larger point attainment signalling better outcome
Change in baseline cognitive function in Trail Making Test (TMT), Parts A & B at 3 months | baseline to 3 months
  The TMT is a validated measure of cognitive function, the time upon completion is measured
Change in baseline cognitive function in Trail Making Test (TMT), Parts A & B at 6 months | baseline to 6 months
  The TMT is a validated measure of cognitive function, the time upon completion is measured
Change in 3 month cognitive function in Trail Making Test (TMT), Parts A & B at 6 months | 3 months to 6 months
  The TMT is a validated measure of cognitive function, the time upon completion is measured
Change in 6 month cognitive function in Trail Making Test (TMT), Parts A & B at 9 months | 6 months to 9 months
  The TMT is a validated measure of cognitive function, the time upon completion is measured
Difference cognitive function in Trail Making Test (TMT), Parts A & B at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  The TMT is a validated measure of cognitive function, the time upon completion is measured
Difference cognitive function in Trail Making Test (TMT), Parts A & B at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  The TMT is a validated measure of cognitive function, the time upon completion is measured
Change in baseline mood in Geriatric Depression Scale at 3 months. | baseline to 3 months
  A self-report measure of mood, measured on 0-15 point scale, higher point attainment signifies worse outcome
Change in baseline mood in Geriatric Depression Scale at 6 months. | baseline to 6 months
  A self-report measure of mood, measured on 0-15 point scale, higher point attainment signifies worse outcome
Change in 3 month mood in Geriatric Depression Scale at 6 months. | 3 months to 6 months
  A self-report measure of mood, measured on 0-15 point scale, higher point attainment signifies worse outcome
Change in 6 month mood in Geriatric Depression Scale at 9 months. | 6 months to 9 months
  A self-report measure of mood, measured on 0-15 point scale, higher point attainment signifies worse outcome
Difference in mood in Geriatric Depression Scale at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  A self-report measure of mood, measured on 0-15 point scale, higher point attainment signifies worse outcome
Difference in mood in Geriatric Depression Scale at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  A self-report measure of mood, measured on 0-15 point scale, higher point attainment signifies worse outcome
Change from baseline self-sufficiency self-reported in Questionnaire of functional state (abbreviation in original language: subjective FAQ-CZ) at 3 months | baseline to 3 months
  FAQ-CZ is a self-report measure of self-sufficiency, it is measured on a scale of 0-30 with higher point attainment signalling worse outcome
Change from baseline self-sufficiency self-reported in Questionnaire of functional state (abbreviation in original language: subjective FAQ-CZ) at 6 months | baseline to 6 months
  FAQ-CZ is a self-report measure of self-sufficiency, it is measured on a scale of 0-30 with higher point attainment signalling worse outcome
Change from 3 month self-sufficiency self-reported in Questionnaire of functional state (abbreviation in original language: subjective FAQ-CZ) at 6 months | 3 months to 6 months
  FAQ-CZ is a self-report measure of self-sufficiency, it is measured on a scale of 0-30 with higher point attainment signalling worse outcome
Change from 6 month self-sufficiency self-reported in Questionnaire of functional state (abbreviation in original language: subjective FAQ-CZ) at 9 months | 6 months to 9 months
  FAQ-CZ is a self-report measure of self-sufficiency, it is measured on a scale of 0-30 with higher point attainment signalling worse outcome
Difference in self-sufficiency self-reported in Questionnaire of functional state (abbreviation in original language: subjective FAQ-CZ) at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  FAQ-CZ is a self-report measure of self-sufficiency, it is measured on a scale of 0-30 with higher point attainment signalling worse outcome
Difference in self-sufficiency self-reported in Questionnaire of functional state (abbreviation in original language: subjective FAQ-CZ) at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  FAQ-CZ is a self-report measure of self-sufficiency, it is measured on a scale of 0-30 with higher point attainment signalling worse outcome
Changes in tau protein | baseline to 3 months
  Measured in pg/ml; 2x10ml samples collected to assess tau protein, neurofilament light and immunocomplex antibody levels
Changes in tau protein | baseline to 6 months
  Measured in pg/ml; 2x10ml samples collected to assess tau protein, neurofilament light and immunocomplex antibody levels
Changes in tau protein | 3 months to 6 months
  Measured in pg/ml; 2x10ml samples collected to assess tau protein, neurofilament light and immunocomplex antibody levels
Changes in tau protein | 6 months to 9 months
  Measured in pg/ml; 2x10ml samples collected to assess tau protein, neurofilament light and immunocomplex antibody levels
Changes in neurofilament light levels | baseline to 3 months
  Measured in pg/ml; 2x10ml samples collected to assess tau protein, neurofilament light and immunocomplex antibody levels
Changes in neurofilament light levels | baseline to 6 months
  Measured in pg/ml; 2x10ml samples collected to assess tau protein, neurofilament light and immunocomplex antibody levels
Changes in neurofilament light levels | 3 months to 6 months
  Measured in pg/ml; 2x10ml samples collected to assess tau protein, neurofilament light and immunocomplex antibody levels
Changes in neurofilament light levels | 6 months to 9 months
  Measured in pg/ml; 2x10ml samples collected to assess tau protein, neurofilament light and immunocomplex antibody levels
Changes in immunocomplex antibody levels | baseline to 3 months
  Measured in ng/ml; 2x10ml samples collected to assess tau protein, neurofilament light and immunocomplex antibody levels
Changes in immunocomplex antibody levels | baseline to 6 months
  Measured in ng/ml; 2x10ml samples collected to assess tau protein, neurofilament light and immunocomplex antibody levels
Changes in immunocomplex antibody levels | 3 months to 6 months
  Measured in ng/ml; 2x10ml samples collected to assess tau protein, neurofilament light and immunocomplex antibody levels
Changes in immunocomplex antibody levels | 6 months to 9 months
  Measured in ng/ml; 2x10ml samples collected to assess tau protein, neurofilament light and immunocomplex antibody levels
Biochemical parameters in blood | baseline to 3 months
  Change from baseline Blood metabolome assessed using mass spectrometry at 3 months
Biochemical parameters in blood | baseline to 6 months
  Change from baseline Blood metabolome assessed using mass spectrometry at 6 months
Biochemical parameters in blood | 3 months to 6 months
  Change from 3 months Blood metabolome assessed using mass spectrometry at 6 months
Biochemical parameters in blood | 6 months to 9 months
  Change from 3 months Blood metabolome assessed using mass spectrometry at 6 months
Biochemical parameters in urine | baseline to 3 months
  15ml sample collected twice at each visitation time point (at home in the morning, during centre visit); Change from baseline Urine metabolome assessed using mass spectrometry at 3 months
Biochemical parameters in urine | baseline to 6 months
  15ml sample collected twice at each visitation time point (at home in the morning, during centre visit); Change from baseline Urine metabolome assessed using mass spectrometry at 6 months
Biochemical parameters in urine | 3 months to 6 months
  15ml sample collected twice at each visitation time point (at home in the morning, during centre visit); Change from 3 months Urine metabolome assessed using mass spectrometry at 6 months
Biochemical parameters in urine | 6 months to 9 months
  15ml sample collected twice at each visitation time point (at home in the morning, during centre visit); Change from 3 months Urine metabolome assessed using mass spectrometry at 6 months
Biochemical parameters in stool | baseline to 3 months
  Change from baseline Stool metabolome assessed using mass spectrometry at 3 months
Biochemical parameters in stool | baseline to 6 months
  Change from baseline Stool metabolome assessed using mass spectrometry at 6 months
Biochemical parameters in stool | 3 months to 6 months
  Change from 3 months Stool metabolome assessed using mass spectrometry at 6 months
Biochemical parameters in stool | 6 months to 9 months
  Change from 3 months Stool metabolome assessed using mass spectrometry at 6 months

SECONDARY OUTCOMES:
Change from baseline Questionnaire of adverse events (abbreviation in original language: DNU) at 3 months | baseline to 3 months
  DNU is a self-report measure of adverse events, scale ranges from 0-22 points with higher point outcome indicating more adverse events
Change from baseline Questionnaire of adverse events (abbreviation in original language: DNU) at 6 months | baseline to 6 months
  DNU is a self-report measure of adverse events, scale ranges from 0-22 points with higher point outcome indicating more adverse events
Change from 3 months Questionnaire of adverse events (abbreviation in original language: DNU) at 6 months | 3 months to 6 months
  DNU is a self-report measure of adverse events, scale ranges from 0-22 points with higher point outcome indicating more adverse events
Change from 6 months Questionnaire of adverse events (abbreviation in original language: DNU) at 9 months | 6 months to 9 months
  DNU is a self-report measure of adverse events, scale ranges from 0-22 points with higher point outcome indicating more adverse events
Difference in the Questionnaire of adverse events (abbreviation in original language: DNU) at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  DNU is a self-report measure of adverse events, scale ranges from 0-22 points with higher point outcome indicating more adverse events
Difference in the Questionnaire of adverse events (abbreviation in original language: DNU) at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  DNU is a self-report measure of adverse events, scale ranges from 0-22 points with higher point outcome indicating more adverse events
Change from baseline Self-assessment of memory at 3 months | baseline to 3 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from baseline Self-assessment of memory at 6 months | baseline to 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from 3 months Self-assessment of memory at 6 months | 3 months to 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from 6 months Self-assessment of memory at 9 months | 6 months to 9 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Difference in Self-assessment of memory at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Difference in Self-assessment of memory at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from baseline Self-assessment of digestion at 3 months | baseline to 3 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from baseline Self-assessment of digestion at 6 months | baseline to 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from 3 months Self-assessment of digestion at 6 months | 3 months to 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from 6 months Self-assessment of digestion at 9 months | 6 months to 9 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Difference in Self-assessment of digestion at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Difference in Self-assessment of digestion at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from baseline Self-assessment of overall health at 3 months | baseline to 3 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from baseline Self-assessment of overall health at 6 months | baseline to 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from 3 months Self-assessment of overall health at 6 months | 3 months to 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from 6 months Self-assessment of overall health at 9 months | 6 months to 9 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Difference in Self-assessment of overall health at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Difference in Self-assessment of overall health at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from baseline Self-assessment of sleep quality at 3 months | baseline to 3 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from baseline Self-assessment of sleep quality at 6 months | baseline to 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from 3 months Self-assessment of sleep quality at 6 months | 3 months to 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from 6 months Self-assessment of sleep quality at 9 months | 6 months to 9 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Difference in Self-assessment of sleep quality at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Difference in Self-assessment of sleep quality at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from baseline Self-assessment of anxiety at 3 months | baseline to 3 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling worse outcome
Change from baseline Self-assessment of anxiety at 6 months | baseline to 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling worse outcome
Change from 3 months Self-assessment of anxiety at 6 months | 3 months to 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling worse outcome
Change from 6 months Self-assessment of anxiety at 9 months | 6 months to 9 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling worse outcome
Difference in Self-assessment of anxiety at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling worse outcome
Difference in Self-assessment of anxiety at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling worse outcome
Change from baseline Self-assessment of fatigue at 3 months | baseline to 3 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling worse outcome
Change from baseline Self-assessment of fatigue at 6 months | baseline to 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling worse outcome
Change from 3 months Self-assessment of fatigue at 6 months | 3 months to 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling worse outcome
Change from 6 months Self-assessment of fatigue at 9 months | 6 months to 9 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling worse outcome
Difference in Self-assessment of fatigue at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling worse outcome
Difference in Self-assessment of fatigue at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling worse outcome
Change from baseline Self-assessment of pain at 3 months | baseline to 3 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from baseline Self-assessment of pain at 6 months | baseline to 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from 3 months Self-assessment of pain at 6 months | 3 months to 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from 6 months Self-assessment of pain at 9 months | 6 months to 9 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Difference in Self-assessment of pain at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Difference in Self-assessment of pain at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  Self-reported on a visual scale ranging from 1-10 with higher point attainment signalling better outcome
Change from baseline physical condition assessment in 30 second sit stand test at 3 months | baseline to 3 months
  Number of sits and stands during 30 seconds
Change from baseline physical condition assessment in 30 second sit stand test at 6 months | baseline to 6 months
  Number of sits and stands during 30 seconds
Change from 3 months physical condition assessment in 30 second sit stand test at 6 months | 3 months to 6 months
  Number of sits and stands during 30 seconds
Change from 6 months physical condition assessment in 30 second sit stand test at 9 months | 6 months to 9 months
  Number of sits and stands during 30 seconds
Difference in physical condition assessment in 30 second sit stand test at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  Number of sits and stands during 30 seconds
Difference in physical condition assessment in 30 second sit stand test at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  Number of sits and stands during 30 seconds
Change from baseline physical condition assessment in 30 second dumbell lift tests at 3 months | baseline to 3 months
  Number lifts during 30 seconds
Change from baseline physical condition assessment in 30 second dumbell lift tests at 6 months | baseline to 6 months
  Number lifts during 30 seconds
Change from 3 months physical condition assessment in 30 second dumbell lift tests at 6 months | 3 months to 6 months
  Number lifts during 30 seconds
Change from 6 months physical condition assessment in 30 second dumbell lift tests at 9 months | 6 months to 9 months
  Number lifts during 30 seconds
Difference in physical condition assessment in 30 second dumbell lift tests at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  Number lifts during 30 seconds
Difference in physical condition assessment in 30 second dumbell lift tests at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  Number lifts during 30 seconds
Change from baseline physical condition assessment in 30 meters walk at 3 months | baseline to 3 months
  Time untill completion
Change from baseline physical condition assessment in 30 meters walk at 6 months | baseline to 6 months
  Time untill completion
Change from 3 months physical condition assessment in 30 meters walk at 6 months | 3 months to 6 months
  Time untill completion
Change from 6 months physical condition assessment in 30 meters walk at 9 months | 6 months to 9 months
  Time untill completion
Difference in physical condition assessment in 30 meters walk at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  Time untill completion
Difference in physical condition assessment in 30 meters walk at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  Time untill completion
Change from baseline Structured nutritional questionnaire about long-term eating habits (abbreviation in original language: STRADO) at 3 months | baseline to 3 months
  Structured self-report questionnaire
Change from baseline Structured nutritional questionnaire about long-term eating habits (abbreviation in original language: STRADO) at 6 months | baseline to 6 months
  Structured self-report questionnaire
Change from 3 months Structured nutritional questionnaire about long-term eating habits (abbreviation in original language: STRADO) at 6 months | 3 months to 6 months
  Structured self-report questionnaire
Change from 6 months Structured nutritional questionnaire about long-term eating habits (abbreviation in original language: STRADO) at 9 months | 6 months to 9 months
  Structured self-report questionnaire
Difference in Structured nutritional questionnaire about long-term eating habits (abbreviation in original language: STRADO) at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  Structured self-report questionnaire
Difference in Structured nutritional questionnaire about long-term eating habits (abbreviation in original language: STRADO) at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  Structured self-report questionnaire
Change in baseline Beck's Anxienty Inventory at 3 months | baseline to 3 months
  Beck's Anxenty Inventory is a validated self-report measure of anxiety. The scale ranges from 0-63 points, higher point attainment signals worse outcome
Change in baseline Beck's Anxienty Inventory at 6 months | baseline to 6 months
  Beck's Anxenty Inventory is a validated self-report measure of anxiety. The scale ranges from 0-63 points, higher point attainment signals worse outcome
Change in 3 months Beck's Anxienty Inventory at 6 months | 3 months to 6 months
  Beck's Anxenty Inventory is a validated self-report measure of anxiety. The scale ranges from 0-63 points, higher point attainment signals worse outcome
Change in 6 months Beck's Anxienty Inventory at 9 months | 6 months to 9 months
  Beck's Anxenty Inventory is a validated self-report measure of anxiety. The scale ranges from 0-63 points, higher point attainment signals worse outcome
Difference in Beck's Anxienty Inventory at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  Beck's Anxenty Inventory is a validated self-report measure of anxiety. The scale ranges from 0-63 points, higher point attainment signals worse outcome
Difference in Beck's Anxienty Inventory (BAI) at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  Beck's Anxenty Inventory is a validated self-report measure of anxiety. The scale ranges from 0-63 points, higher point attainment signals worse outcome
Change in baseline Beck's Depression Inventory - II (BDI-II) at 3 months | baseline to 3 months
  BDI-II is a validated self-report measure of depression with scale ranging from 0-63 points, higher point attainment signals worse outcome
Change in baseline Beck's Depression Inventory - II (BDI-II) at 6 months | baseline to 6 months
  BDI-II is a validated self-report measure of depression with scale ranging from 0-63 points, higher point attainment signals worse outcome
Change in 3 months Beck's Depression Inventory - II (BDI-II) at 6 months | 3 months to 6 months
  BDI-II is a validated self-report measure of depression with scale ranging from 0-63 points, higher point attainment signals worse outcome
Change in 6 months Beck's Depression Inventory - II (BDI-II) at 9 months | 6 months to 9 months
  BDI-II is a validated self-report measure of depression with scale ranging from 0-63 points, higher point attainment signals worse outcome
Difference in Beck's Depression Inventory - II (BDI-II) at 3 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 3 months
  BDI-II is a validated self-report measure of depression with scale ranging from 0-63 points, higher point attainment signals worse outcome
Difference in Beck's Depression Inventory - II (BDI-II) at 6 months between the Probiotics C2P/Placebo and Placebo/C2P Probiotics group | 6 months
  BDI-II is a validated self-report measure of depression with scale ranging from 0-63 points, higher point attainment signals worse outcome

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - University Hospital Vinohrady, Prague
  - National Institute of Mental Health, Czech Republic, Prague

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Bartos A, Weinerova J, Diondet S. Effects of human probiotics on memory and psychological and physical measures in community-dwelling older adults with normal and mildly impaired cognition: results of a bi-center, double-blind, randomized, and placebo-controlled clinical trial (CleverAge biota). Front Aging Neurosci. 2023 Jul 7;15:1163727. doi: 10.3389/fnagi.2023.1163727. eCollection 2023. PMID 37502424
- [Derived] Bartos A, Weinerova J, Diondet S, Vales K. Effect of human probiotics on memory, psychological and biological measures in elderly: A study protocol of bi-center, double-blind, randomized, placebo-controlled clinical trial (CleverAge Biota). Front Aging Neurosci. 2022 Nov 10;14:996234. doi: 10.3389/fnagi.2022.996234. eCollection 2022. PMID 36437993
- See also: National Institute of Mental Health - official website — https://www.nudz.cz/en/